CLINICAL TRIAL: NCT01875874
Title: An Open-Label, Multicenter, Historically-Controlled Study to Assess Safety and Efficacy of ELAD in Subjects With Acute Liver Failure (ALF)
Brief Title: Safety and Efficacy of the ELAD System (ELAD) to Treat Acute Liver Failure (ALF)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to VTI-208 results, the ELAD clinical plan is being re-evaluated.
Sponsor: Vital Therapies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VTI-212
Record Dates: First submitted 2013-06-05; First posted 2013-06-12 (Estimated); Results first posted 2018-08-22 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-01

CONDITIONS: Acute Liver Failure; Fulminant Hepatic Failure; Primary Graft Non-Function; Surgically-Induced Liver Failure
Keywords: liver failure; acute liver failure; fulminant hepatic failure; primary graft non-function; surgically-induced liver failure; ELAD; ALF; FHF; PNF
MeSH Terms: conditions — Liver Failure, Acute; Liver Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ELAD plus standard of care (Experimental): Continuous ELAD treatment for a minimum of 3 days to a maximum of 10 days in addition to a standard of care for subjects with acute liver failure.
  Interventions: Biological: ELAD

INTERVENTIONS:
Biological: ELAD — Continuous treatment with the ELAD System for a minimum of 3 days to a maximum of 10 days. The subject's ultrafiltrated blood is circulated through 4 cartridges, each containing approximately 110 grams of C3A cells (approximately 440 grams total).
  Other Names: Human Cell-Based Bio-Artificial Liver Support System

SUMMARY:
This phase 2 study is developed to evaluate the effect of ELAD on overall survival (OS) in subjects with acute liver failure (ALF) compared to matched historical controls.

DETAILED DESCRIPTION:
The VTI-212 study (VTI-212) is an open-label, multicenter, historically-controlled study of subjects with acute liver failure (ALF). Approximately 40 subjects who meet the eligibility requirements of the study will receive ELAD treatment in addition to standard of care treatment for ALF. The outcomes of these subjects will be compared with matched historical controls drawn from existing databases.

Subjects will undergo ELAD treatment for a minimum of 3 days (72 hours). It is recommended ELAD treatment be continued up to 10 days (240 hours).

Following ELAD treatment, subjects will continue standard medical therapy as defined by the institution and be followed through Study Day 28.

Subjects' diagnosis of ALF will be attributed to one of the following:

1. Fulminant Hepatic Failure (FHF) (acute liver failure with no preexisting liver disease);
2. Primary Graft Non-Function (PNF);
3. Surgically-Induced Liver Failure (including subjects with small for size liver transplants, living donor liver transplants, and subjects with risk of ALF following liver cancer surgery.

Screening evaluations and assessments will be completed for subjects and reviewed against inclusion/exclusion criteria.

Enrollment will define the time of study entry (Hour 0, Study Day 1, study baseline) and inclusion in the Intent-to-treat (ITT) population. Subjects will be evaluated throughout the 28-day study period.

If standard medical therapy, as defined by the institution and this protocol is consistent with discharging the subject home, then the subject should be discharged. Prior to discharge, the subject will be advised to attend all follow-up visits.

An extension of this study, the VTI-212E study (VTI-212E), will provide additional ELAD survival data, as available, through VTI-212 study termination (after the last surviving enrolled ELAD subject completes Study Day 28). This registry protocol segment of VTI-212 extends the safety monitoring period to 5 years to assess survival, incidence and characterization of tumor (in particular hepatocellular tumor), incidence of liver transplant, and assess quality of life using a standard, validated questionnaire.

The ITT population includes all randomized subjects assigned to the group to which they were randomized, irrespective of actual treatment administered. Participant, Baseline Characteristics, and Outcome Measures used the ITT population. The safety population is defined as all subjects who are randomized based on actual treatment received. All serious adverse events and all non-serious adverse events analyses used the safety population.

ELIGIBILITY:
Inclusion Criteria:

1. Weight ≥ 40 kg;
2. Age ≥ 18;
3. Diagnosis of ALF attributed to one of the following:

   1. FHF (acute liver failure with no preexisting liver disease, see below);
   2. Primary Graft Non-Function (PNF);
   3. Surgically-Induced Liver Failure (including subjects with small for size liver transplants, living donor liver transplants, and subjects with risk of ALF following liver cancer surgery);
4. Subjects must not be listed for transplant at the time of Enrollment or, if listed, in the opinion of the Investigator are unlikely to be transplanted within 72 hours;
5. Subject or legally authorized representative must provide Informed Consent for VTI-212 and the Follow-up Registry VTI-212E.

   Subjects with FHF must meet one of the following criteria:
6. Known acetaminophen ingestion or diagnostic serum level, and at least one of the following:

   1. Prothrombin time (PT) > 100 seconds [International Normalized Ratio (INR) > 6.5], OR
   2. Encephalopathy Grade 3 or 4 AND ARTERIAL AMMONIA >100 umol/liter and at least one of the following:

   i. Arterial pH < 7.30 at ≥ 24 hours after drug ingestion or volume resuscitation; ii. Renal failure documented by urine output < 0.5 mL/kg/hr over the preceding 12 hours; iii. Creatinine > 2.5 mg/dL; OR
7. Non-acetaminophen-induced FHF with Encephalopathy Grade 3 or 4 and arterial ammonia >100 umol/liter, and at least two of the following:

   1. Viral Hepatitis (other than A, B or C) or drug (non-acetaminophen)-induced FHF
   2. Serum bilirubin > 17 mg/dL
   3. Subject > 40 years old
   4. PT > 50 seconds (INR > 3.5)
   5. Jaundice to encephalopathy time ≥ 7 days

Exclusion Criteria:

1. Cerebral Perfusion Pressure ≤40 mm Hg for 1 hour or longer as measured by an intracranial pressure (ICP) monitor. (NOTE: In those cases where ICP monitor placement cannot be performed prior to study enrollment, this exclusion criterion will not apply);
2. Chronic liver disease (e.g., compensated cirrhosis of any etiology, chronic hepatitis, nonalcoholic steatohepatitis, cholestatic liver disease, or metabolic liver disease) (NOTE: steatosis is not an exclusion criterion);
3. Acute clinical symptoms that, in the Investigator's opinion, are likely to result in death within 48 hours of enrollment;
4. Evidence of infection unresponsive to antibiotics (e.g. increased tissue involvement relative to initial diagnosis, clinical worsening of symptom) indicated by any of the following:

   1. Presence of sepsis or septic shock; OR
   2. Positive blood cultures (bacteremia, fungemia) within 72 hours prior to Enrollment; OR
   3. Presence of spontaneous bacterial peritonitis during the 2 days prior to Enrollment; OR
   4. Clinical and radiological signs of pneumonia.
5. Concomitant disease including chronic congestive heart failure, severe vascular disease, emphysema, AIDS, cancer (except non-melanoma skin cancer), acute fatty-liver disease, hepatitis due to herpes virus or Budd-Chiari syndrome. (NOTE: in the case of subjects enrolled due to surgery-induced liver failure (SILF) then the original cause for the surgery will not be a criterion for exclusion);
6. Portal hypertension;
7. Liver dysfunction due to trauma;
8. Irreversible brain death;
9. Platelet count < 30,000/mm3 [NOTE: Subject may be included at the physician's discretion if platelet count exceeds 30,000/mm3 at time of initiation of therapy (even if the value is following platelet transfusion) and can be managed through the administration of blood products]
10. Cardiovascular sepsis-related organ failure assessment score (SOFA score) >3;
11. Stroke or intracranial hemorrhage;
12. Seizures uncontrolled by medication;
13. Acute myocardial infarction;
14. Lung disease defined by a partial pressure of oxygen measurement (PaO2) ≤60 mmHg or a fraction of inspired oxygen (FiO2) ≥0.6, not corrected by medical management [including continuous venovenous hemofiltration (CVVH) if indicated] and ventilation with a Positive End Expiratory Pressure (PEEP) of >8cm H2O;
15. Acute Respiratory Distress Syndrome;
16. Pregnancy as determined by beta-human chorionic gonadotropin (β-hCG) results;
17. ≤ 2 weeks postpartum;
18. Participation in another investigational drug, biologic, or device study within one month of enrollment, except for observational studies (the observational study setting should not affect the safety and/or efficacy of the VTI-212 clinical trial);
19. Prior ELAD therapy;
20. Has a Do Not Resuscitate or a Do Not Intubate (DNR/DNI) directive (or local equivalent) or any other Advanced Directive limiting Standard of Care in place (the DNR/DNI criterion is not applicable in the UK).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-10; Primary Completion 2015-09 (Actual); Study Completion 2018-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Stange, MD, Ph.D., Study Chair — Vital Therapies, Inc.; Parvez Mantry, MD, Principal Investigator — TX - Methodist Dallas Medical Center - The Liver Institute; David J Reich, MD, Principal Investigator — PA - Drexel University College of Medicine; Paul J Gaglio, MD, Principal Investigator — NY - Montefiore Medical Center; Juan Gallegos-Orozco, MD, Principal Investigator — UT - University of Utah; Angel Alsina, MD, Principal Investigator — FL - Tampa General Hospital; Lewis W Teperman, MD, Principal Investigator — NY - New York University Medical Center; Nikunj Shah, MD, Principal Investigator — IL - Rush University Medical Center; Julie Thompson, MD, Principal Investigator — MN - University of Minnesota Medical Center - Twin Cities Campus; Winfred W Williams, Jr., MD, Principal Investigator — MA - Massachusetts General Hospital; Lance Stein, MD, Principal Investigator — GA - Piedmont Atlanta Hospital; Ram Subramanian, MD, Principal Investigator — GA - Emory University Hospital; Nikolaos T Pyrsopoulos, MD, Principal Investigator — NJ - Rutgers University Hospital; Marquis Hart, MD, Principal Investigator — WA - Swedish Medical Center; Rohit Satoskar, MD, Principal Investigator — DC - Georgetown University Hospital; Talal Adhami, MD, Principal Investigator — OH - Cleveland Clinic Foundation; Linda S Sher, MD, Principal Investigator — CA - Keck Hospital of USC; Xaralambos Zervos, DO, Principal Investigator — FL - Cleveland Clinic Florida; Kalyan R Bhamidimarri, MD, Principal Investigator — FL - University of Miami Hospital
Locations (18):
- United States (18):
  - Keck Hospital of USC, Los Angeles, California
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - University of Miami Hospital, Miami, Florida
  - Tampa General Hospital, Tampa, Florida
  - Cleveland Clinic Floriday, Weston, Florida
  - Piedmont Atlanta Hospital, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Minnesota Medical Center - Twin Cities Campus, Minneapolis, Minnesota
  - Rutgers University Hospital, Newark, New Jersey
  - New York University Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - Methodist Dallas Medical Center - The Liver Institute, Dallas, Texas
  - University of Utah, Salt Lake City, Utah
  - Swedish Medical Center, Seattle, Washington

REFERENCES:
- See also: Vital Therapies, Inc. website — http://www.vitaltherapies.com

RESULTS

PARTICIPANT FLOW:
Groups:
- ELAD System (ELAD) Treatment Plus Standard of Care Treatment: Continuous treatment with the ELAD System (ELAD) for a minimum of 3 days to a maximum of 10 days in addition to a standard of care for subjects with acute liver failure.
  ELAD: Continuous treatment with the ELAD System for a minimum of 3 days to a maximum of 10 days. The subject's ultrafiltrated blood is circulated through 4 cartridges, each containing approximately 110 grams of C3A cells (approximately 440 grams total).
Period: Overall Study
Arm/Group | ELAD System (ELAD) Treatment Plus Standard of Care Treatment
Started | 8
Completed | 5
Not Completed | 3
Not completed — Death | 3

BASELINE CHARACTERISTICS:
Population: Same phrase as in AE section.
Groups:
- ELAD Treatment Plus Standard of Care Treatment: Continuous ELAD treatment for a minimum of 3 days to a maximum of 10 days in addition to a standard of care for subjects with acute liver failure.
  ELAD: Continuous treatment with the ELAD System for a minimum of 3 days to a maximum of 10 days. The subject's ultrafiltrated blood is circulated through 4 cartridges, each containing approximately 110 grams of C3A cells (approximately 440 grams total).
Arm/Group | ELAD Treatment Plus Standard of Care Treatment
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.5 (19.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) of ALF Subjects
Time Frame: Study Day 1 through Study Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | ELAD Treatment Plus Standard of Care Treatment
Number analyzed (Participants) | 8
Participants | 5

2. Secondary Outcome: Number of Subjects Who Survived at the End of Study Day 28 or Who Received Orthotopic Liver Transplantation on or Before That Study Day.
Time Frame: Study Day 1 through Study Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | ELAD System (ELAD) Treatment Plus Standard of Care Treatment
Number analyzed (Participants) | 8
Participants | 5

ADVERSE EVENTS:
Description: One subject was not treated with ELAD due to substantial improvement of their condition prior to treatment initiation. Therefore, only 7 subjects were exposed to ELAD treatment and at risk for adverse events.
Arm/Group | ELAD Treatment Plus Standard of Care Treatment
All-Cause Mortality (participants affected / at risk) | 3/7
Serious Adverse Events (participants affected / at risk) | 6/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ELAD Treatment Plus Standard of Care Treatment (N=7)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Multi-organ failure (General disorders) | 3 (3)
Autoimmune hepatitis (Hepatobiliary disorders) | 1 (1)
Liver transplant rejection (Immune system disorders) | 1 (2)
Hyperammonaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ELAD Treatment Plus Standard of Care Treatment (N=7)
Anaemia (Blood and lymphatic system disorders) | 5 (6)
Anaemia macrocytic (Blood and lymphatic system disorders) | 1 (1)
Hypofibrinogenaemia (Blood and lymphatic system disorders) | 2 (2)
Leukocytosis (Blood and lymphatic system disorders) | 3 (3)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
Arrhythmia supraventricular (Cardiac disorders) | 1 (1)
Cyanosis (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 4 (4)
Ventricular arrhythmia (Cardiac disorders) | 1 (1)
Dry eye (Eye disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Oral mucosa erosion (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Application site necrosis (General disorders) | 1 (1)
Catheter site haematoma (General disorders) | 1 (1)
Catheter site haemorrhage (General disorders) | 3 (3)
Chest pain (General disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Gait disturbance (General disorders) | 1 (1)
Generalized oedema (General disorders) | 1 (1)
Hypothermia (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 2 (2)
Pain (General disorders) | 1 (1)
Peripheral swelling (General disorders) | 1 (1)
Pyrexia (General disorders) | 4 (5)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1)
Biliary fistula (Hepatobiliary disorders) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (3)
Sepsis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Complications of transplant surgery (Injury, poisoning and procedural complications) | 2 (2)
Hepatic haematoma (Injury, poisoning and procedural complications) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (1)
Alpha 1 foetoprotein increased (Investigations) | 1 (1)
Amylase increased (Investigations) | 1 (1)
Body temperature increased (Investigations) | 1 (1)
Candida test positive (Investigations) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 1 (1)
Electrocardiogram ST segment elevation (Investigations) | 1 (1)
Electrocardiogram T wave inversion (Investigations) | 1 (1)
Liver function test abnormal (Investigations) | 1 (1)
Occult blood positive (Investigations) | 2 (2)
Oxygen saturation decreased (Investigations) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 1 (1)
Hyperammonaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2)
Hypermagnesaemia (Metabolism and nutrition disorders) | 2 (2)
Hyperphosphataemia (Metabolism and nutrition disorders) | 2 (2)
Hypervolaemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hypochloraemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Brain injury (Nervous system disorders) | 1 (1)
Intracranial pressure increased (Nervous system disorders) | 1 (1)
Agitation (Psychiatric disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 4 (5)

LIMITATIONS AND CAVEATS:
This study was terminated early, after enrollment of only 8 out of 40 planned subjects, due to findings from previous VTI-208 study. Thus, sample size of VTI-212 was very small leading to statistical analyses that cannot be meaningfully interpreted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes